CLINICAL TRIAL: NCT00460954
Title: An Open Label, Multiple-Dose Study ot Determine the Plasma Levodopa Profiles of Sinemet® CR (Carbidopa/Levodopa) at 4 Daily Dose Levels in Healthy Subjects
Brief Title: A Multiple-Dose Study of Sinemet® CR (Carbidopa/Levodopa) in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Other Study IDs: CN158-001
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Carbidopa; Levodopa

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Sinemet® controlled release (Carbidopa/levodopa)

SUMMARY:
The purpose of this clinical research study is to determine if different dosage regimens of Sinemet® CR (Carbidopa/levodopa) are dose proportional

ELIGIBILITY:
* Key inclusion and exclusion criteria for healthy volunteers will be used
* Males and females aged 50-75

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-06; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Toronto, Ontario, Canada